CLINICAL TRIAL: NCT00536692
Title: Phase 2 Study of the Safety and Bioactivity of Topical Ocular Mecamylamine for the Treatment of Diabetic Macular Edema (DME)
Brief Title: Topical Ocular Mecamylamine in Diabetic Macular Edema (DME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CoMentis (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG003-202
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Diabetic Macular Edema
Keywords: macular edema; DME; diabetic; mecamylamine; Comentis
MeSH Terms: conditions — Macular Edema | interventions — Mecamylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mecamylamine — topical ocular drops

SUMMARY:
This is an open-label study evaluating the safety and tolerability of topical ocular mecamylamine given twice a day in patients with diabetic macular edema (DME). Patients will be treated for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* macular edema due to diabetic retinopathy

Exclusion Criteria:

* vision loss from other ocular disease
* intraocular surgery within 3 months
* intraocular anti-VEGF or steroids within 3 months
* HbA1c >12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - East Bay Retina Consultants, Inc., Oakland, California
  - Johns Hopkins School of Medicine / Wilmer Eye Institute, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts

REFERENCES:
- [Derived] Campochiaro PA, Shah SM, Hafiz G, Heier JS, Lit ES, Zimmer-Galler I, Channa R, Nguyen QD, Syed B, Do DV, Lu L, Monk J, Cooke JP, Kengatharan MK, Hsu HH. Topical mecamylamine for diabetic macular edema. Am J Ophthalmol. 2010 May;149(5):839-51.e1. doi: 10.1016/j.ajo.2009.12.005. Epub 2010 Feb 26. PMID 20189159